CLINICAL TRIAL: NCT06029361
Title: Improving Function and Mobility in Geriatric Patients After a Femoral Neck Fracture Who Are Undergoing Inpatient Rehabilitation Using an Augmented Reality Practice System - SELFIT
Brief Title: Improvement of Function After Hip Fracture in Geriatric Rehabilitation Unit Via Augmented Reality Device "SELFIT"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Protsenko, Head of physiotherapy of geriatric rehabilitation unit, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0003-22 MMC
Record Dates: First submitted 2023-08-23; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Control Groups

STUDY DESIGN:
Masking Description: an assessment will be made by questionnaires and an objective assessment by physiotherapists who will not be involved in the treatment of the SELFIT system in the interventional group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SELFIT device group (Experimental): 25 patients in experimental group will receive 15 minutes with the SELFIT system during the 45 minutes of physical therapy
  Interventions: Device: Selfit Device group
- Control Group (Active Comparator): 45 minutes of conventional physical therapy
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Selfit Device group — During 21 days, intervention group will receive physical therapy of 45 minutes which 15 minutes out of the 45 minutes will be with the SELFIT system
  Arms: SELFIT device group
Other: Control Group — Conventional physical therapy of 45 minute
  Arms: Control Group

SUMMARY:
Type of study: prospective interventional the purposes of the research :To examine the effect of treatment using the SELFIT system on function, walking and balance in patients after hip fractures hospitalized in the geriatric rehabilitation department.

The study population: 50 participants aged 65+ who were admitted to the geriatric rehabilitation department after hip fractures, with 25 in the experimental group and 25 in the control group.

The main question[s] it aims to answer are:

* What is the effect of training with SELFIT system on the functional outcomes in patients after hip fractures hospitalized in the geriatric rehabilitation department.
* How the training with SELFIT system will effect on satisfaction of the patients in the geriatric rehabilitation department.

During 21 days, both groups will receive physical therapy for about 45 minutes. The experimental group will be allocated about 15 minutes out of the 45 minutes to practice with the help of the SELFIT system.

DETAILED DESCRIPTION:
Recruiting participants for the study:

When admitting patients hospitalized in the geriatric rehabilitation department after hip neck fractures, their suitability for participation in the study will be examined according to inclusion and exclusion criteria. Patients who meet the inclusion criteria will receive an explanation of the research procedure and its goals, and if they agree and are suitable in terms of signature competence and cognitive ability to participate in the study, they will sign an informed consent form for participation in the study.

After signing a consent form to participate in the study, each participant will be randomly assigned to an experimental group or a control group. After the patient agrees to participate in the study, he will receive a number that will be assigned in sequential order, where an even number means belonging to the experimental group and an odd number, belonging to the control group.

Intervention:

During 21 days, both groups will receive physical therapy for about 45 minutes. The experimental group will be allocated about 15 minutes out of the 45 minutes to practice with the help of the SELFIT system.

Both groups will receive physiotherapy treatment accepted in the geriatric rehabilitation department. Patients in both groups receive treatment that focuses on improving strength in the lower limbs, improving ROM, lying and standing exercises, walking with an assistive device according to the patient's ability.

In the second and third week of rehabilitation, patients progress to exercises to improve walking ability, which include standing practice to improve strength and balance, walking with an aid for distances according to the adjustment of walking ability, dynamic balance practice on unstable surfaces and practice on stairs.

Patients from the control group will receive standard treatment according to the patient's ability and the degrees of difficulty of the exercises will progress according to the ability of each patient. After the evaluation, the patients in the control group will receive an exercise in bed lying down or sitting to strengthen the lower limbs for about 15 minutes, an exercise in front of a bar to improve the strength of the lower limbs and the ability to stand up for about 15 minutes, an exercise to improve balance and walking for about 15 minutes.

Patients from the experimental group will receive exercise in bed lying down or sitting to strengthen lower limbs for about 15 minutes, exercise in front of a bar to improve lower limb strength and the ability to stand up for about 15 minutes, exercise in the SELFIT system of balance and walking for about 15 minutes. The intervention in the SELFIT system will be carried out 4 times a week by a physiotherapist in the department.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk independently or under supervision before the fracture
* Patients with full weight bearing on the operated leg according to the instructions of an orthopedic surgeon (FWB - Full Weight Bearing)
* Patients who are able to walk with an assistive device FIM 3 and above (FIM Functional independence measure)
* Mental competence after a comprehensive assessment by a Geriatric Specialist

Exclusion Criteria:

* Patients with cognitive decline following dementia or delirium
* Patients with complications after surgery - infection or bleeding in the surgical area
* Patients with previous neurological injury or current CNS disease.
* Patients with a previous lower limb fracture in the last 5 years.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure | 9 month
  Measured by: Functional Independence Measure Index (FIM) that assess activity of daily living.
  only motor assessment part is used. Minimum score 5 pts. Maximum score: 35 points.
  Higher score means better outcome
5 time sit to stand | 9 month
  Assessment of time performance for five time stand up and sitting on chair. Less time means better outcome
Berg Balance Test | 9 month
  Assessment of balance function by 14 tasks. Min.0 max.56 points Higher score means better outcome.
10 Meter walk test | 9 month
  Assessment of time performance of walking 10 meters. Less time means better outcome
Falls Efficacy Scale | 9 month
  Assessment of confidence of functions. Score range from 16 to 64 points. Higher score means better outcomes
VAS - visual analog scale | 9 month
  as mesured by a pain scale from 1 to 10. Lower score means better outcome
PTPSQ-H physical therapy satisfaction questionnaire | 9 month
  Hebrew approved version. 15 questions about patient satisfaction with physical therapy care. Score range about 15 to 75.
  Higher score means better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel